CLINICAL TRIAL: NCT02863042
Title: Is Deltoid Ligament Repair in Supination-external Rotation Ankle Fractures Necessary? A Prospective Cohort Study.
Brief Title: Is Deltoid Ligament Repair for Ankle Fracture Necessary?
Acronym: AnkleFX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI pulled the study. No participants.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Glenn G. Shi, M.D., Orthopedic Consultant, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-003179
Record Dates: First submitted 2016-05-19; First posted 2016-08-11 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Deltoid Tendon Repaired (Experimental): Repair Deltoid Tendon
  Interventions: Procedure: Repair Deltoid Tendon
- Ankle Fracture Without Deltoid Tendon Repair (Other)
  Interventions: Other: Ankle Fracture Without Deltoid Tendon Repair

INTERVENTIONS:
Procedure: Repair Deltoid Tendon
  Arms: Deltoid Tendon Repaired
Other: Ankle Fracture Without Deltoid Tendon Repair — Standard of care
  Arms: Ankle Fracture Without Deltoid Tendon Repair

SUMMARY:
The investigator hypothesizes that primary acute ankle deltoid ligament repair can help restore ankle radiographic congruity and functional outcomes.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether stabilization with anatomic ankle deltoid ligament repair can help restore ankle congruity and improve functional outcome in patients with unstable supination-external rotation ankle fractures.

ELIGIBILITY:
Inclusion criteria:

* Supination-external rotation ankle fracture with deltoid ligament incompetency
* Minimum of 2 year clinical follow up

Exclusion criteria:

* Non-supination-external rotation ankle fracture
* Medial malleolus fracture
* Incomplete clinical or radiographic followup.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Change in Functional Improvement as measured by the Short Musculoskeletal Function Assessment (SMFA) | baseline, 6 month post-operative visit
  The 46-item SMFA questionnaire comprises two parts: the dysfunction index with 34 items and the bother index with 12 items. Each item has a 5-point response format (1 point for good function or not bothered and 5 points for poor function or extremely bothered).
  The scores of the dysfunction and the bother indices are calculated by summing up the responses to the items and then transforming the scores according to the formula: (actual raw score - lowest possible raw score)/(possible range of raw score) × 100. This transformation formula gives the final scores, which ranged from 0 to 100. The higher scores indicate poorer function.

SECONDARY OUTCOMES:
Mean Score on American Orthopaedic Foot and Ankle Society (AOFAS) Hindfoot Scale | 2 year postoperative visit
  The AOFAS Hindfoot Scale is an outcome rating system for ankle replacements. It is composed of the parameters pain (max 40 points), function (max 50 points) and alignment (max 10 points). Scores can range from 0 (severe pain, severely impaired function, and poor alignment) to 100 (no pain, no limitations on function, good alignment.)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn G Shi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No